CLINICAL TRIAL: NCT01155245
Title: Study on the Effect of 24 Months of Teriparatide Therapy on Bone Microarchitecture and Bone Volume in Postmenopausal Women With Osteoporosis
Brief Title: Teriparatide (PTH) and Bone Strength in Postmenopausal Women
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 08-0321
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2023-05

CONDITIONS: Osteoporosis
Keywords: osteoporosis; HR-pQCT; PTH
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Forteo (teriparatide): postmenopausal women with osteoporosis
  Interventions: Drug: Forteo
- Forteo (teriparatide) with AFF: Women with atypical femur fractures
  Interventions: Drug: Forteo

INTERVENTIONS:
Drug: Forteo — Forteo pen

SUMMARY:
This study will investigate the effects on bone quality of a medication (Teriparatide) used to treat people with severe osteoporosis. Teriparatide is the only bone formation therapy that has been approved for the treatment of postmenopausal osteoporosis in Canada. Osteoporosis is currently diagnosed using a bone mineral density (BMD) scan, which measures the amount of mineral (calcium etc) in bones (the higher the amount of mineral, the lower the fracture risk). Although BMD is linked to bone strength and is used to measure fracture risk, it does not give information on bone structure (called bone geometry) which can also tell us a great deal about fracture risks. Clinical trials have shown that teriparatide increases BMD at the lumbar spine and total hip, while BMD at the forearm decreases after 20 months of therapy. Whether this decrease of BMD at the forearm suggests a higher risk of wrist fracture or a change in bone structure is unclear. Bone biopsies of the pelvis done on people taking teriparatide shows improvement of bone geometry (ie bone thickness and increased trabeculae (small interconnecting rods of bone), suggesting that a change in bone geometry at the wrist may be occurring as well. Currently, there is a new technology, high resolution pQCT (HR-pQCT) that can assess bone geometry without a biopsy. Since bone strength is affected both by BMD and bone structure (as well as other material properties), our group is interested in examining changes in bone geometry at the forearm (a non-weight bearing site) and ankle (a weight bearing site) in postmenopausal women with osteoporosis who receive 24 months of teriparatide therapy. The investigators believe that this new approach of measuring bone strength will help us better understand whether teriparatide has different effects at different bone sites.

DETAILED DESCRIPTION:
This study will investigate the effects on bone quality of a medication used to treat severe osteoporosis. Teriparatide (PTH) is the only bone formation therapy that has been approved for the treatment of postmenopausal osteoporosis in Canada. It works by inducing new periosteal bone apposition, which results in improved bone geometry and increased bone strength, changes that may not be captured by bone mineral density (BMD) measurements. Randomized controlled trials have shown that teriparatide increases BMD at the lumbar spine and total hip, while BMD at the forearm may decrease after 20 months of therapy. As no data to date has been published on changes in bone geometry at the radius either by bone biopsy or high resolution peripheral quantitative computer tomography (HR-pQCT) in patients receiving PTH therapy, it is unclear whether the decline in BMD at the distal radius observed during PTH therapy is indicative of decreases in bone strength, or is a result of increases in the width of the radius. It is our intention to fill this gap in knowledge with regard to how PTH affects BMD and bone structure at the radius and tibia in postmenopausal women with severe osteoporosis. Examining these two components will enable us to better understand the effect of teriparatide on bone strength at the radius and the tibia, and bone strength in general, independent of changes in BMD after a course of treatment.

The main objectives of this study are to determine the effect of 24 months of teriparatide therapy on cortical thickness, trabecular thickness, trabecular number, trabecular separation and BV/TV, as measured by HR-pQCT (XtremeCT, Scanco Medical, Switzerland) at the radius and tibia in postmenopausal women with osteoporosis. The primary outcome will be cortical thickness; the other measures will be secondary outcomes. The secondary objective is to determine the effect of 24 months of teriparatide therapy on moment of inertia, connectivity index, and bone strength, as measured by the HR-pQCT and calculated using finite element modeling analysis at the radius and tibia in postmenopausal women with osteoporosis.

This is an open label before and after study of a cohort of postmenopausal women taking teriparatide at baseline and at 24 months of teriparatide therapy. Recruitment of these subjects will be by referral from specialty clinics of the participating investigators. The postmenopausal women in this study will be prescribed teriparatide according to the most recent Canadian product monograph for Forteo™. Participants will undergo two(2) procedures on five(5) separate occasions (at baseline, 6 months, 12 months, 18 months and at 24 months). The procedures are HR-pQCT and DEXA. In addition to the above procedures, subjects will be asked to complete blood tests which are part of standard clinical practice. Blood will be drawn both at baseline and at 1 month. A follow up phone call will also be made to the participant at 1, 6, and 12 months to discuss any updates in health status.

With this data, the investigators hope to provide a better understanding of the changes that occur in bone structure at the distal radius and tibia during teriparatide therapy.

ELIGIBILITY:
Inclusion Criteria:

* History of fragility fracture OR
* High risk for fractures OR
* Very low BMD (T-score ≤ -2.5) OR
* Failed or intolerant to bisphosphonates
* Baseline serum levels of calcium, urate, ALP, PTH, creatinine and 25-hydroxyvitamin D [25(OH)D] must be within acceptable normal limits

Exclusion Criteria:

* History of skeletal irradiation
* Those at increased risk for osteosarcoma
* Diagnosis of Paget's disease
* History of primary hyperparathyroidism
* Significant renal impairment
* Vitamin D deficiency
* On steroids or have other causes of secondary osteoporosis

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: community dwelling postmenopausal women with osteoporosis and women with atypical femur fractures
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-06; Primary Completion 2024-01 (Actual); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in cortical thickness with teriparatide therapy from baseline to 24 months | 0 to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Angela MW Cheung, MD, PhD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, TGH, Toronto, Ontario, Canada